CLINICAL TRIAL: NCT07309692
Title: Three Dimensional Ultrasonography Versus Hysteroscopy for the Evaluation of Patients With Perimenopausal Bleeding
Brief Title: Different Modalities for the Evaluation of Patients With Peri-menopausal Bleeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Abd Al Rahim Fattouh, Resident doctor at obstetric and gynecology department of sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-25-9----11MS
Record Dates: First submitted 2025-11-27; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Perimenopausal Bleeding
Keywords: ultrasonography; hysteroscopy
MeSH Terms: interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with perimenopausal bleeding (Experimental)
  Interventions: Diagnostic Test: three dimensional ultrasonography; Diagnostic Test: Hysteroscopy

INTERVENTIONS:
Diagnostic Test: three dimensional ultrasonography — all recruited patients will be subjected to three dimensional ultrasonography to diagnose the cause of perimenopausal bleeding
Diagnostic Test: Hysteroscopy — diagnostic hysteroscopy will be performed to diagnose the cause of perimenopausal bleeding

SUMMARY:
The study aims to compare between 3D ultrasonography and hysteroscopy for the evaluation of cases with Peri-menopausal bleeding

ELIGIBILITY:
Inclusion Criteria:

Any pattern of abnormal uterine bleeding as menorrhagia or metrorrhagia for more than 3 months at age between 40 and 55 years , and no ovarian lesion or local cause of bleeding as vaginal or cervical ulcer

Exclusion Criteria:

* • Women with postmenopausal bleeding.

  * Systemic causes of perimenopausal bleeding DM Hypertension or chronic liver disease.
  * Women on hormonal therapy or using any contraception as IUD.
  * Women have contraindication for hysteroscopy as cervical stenosis or pregnancy.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of the 3D ultrasonography for the diagnosis of the causes of peri-menopausal bleeding as compared to hysteroscopy | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dokara-Friedrich ML, Loeffler M, Shehaj I, Tahmasbi-Rad M, Gasimli B, Karn T, Sanhaji M, Becker S, Gasimli K. The Clinical Relevance of Fractional Curettage in the Diagnostic Management of Primary Endometrial Cancer. Gynecol Obstet Invest. 2024;89(4):311-322. doi: 10.1159/000538268. Epub 2024 Mar 12. PMID 38471484
- [Result] Saponara S, Angioni S, Parry JP, Pacheco LA, Carugno J, Moawad N, Haimovich S, Lasmar RB, Dealberti D, Aksakal E, Urman B, Nappi L, Vitale SG. The Pivotal role of hysteroscopy in diagnosing subtle uterine lesions in infertile patients: Seeing the unseen can make the difference. Eur J Obstet Gynecol Reprod Biol. 2025 Feb;305:132-141. doi: 10.1016/j.ejogrb.2024.12.013. Epub 2024 Dec 9. PMID 39701007
- [Result] Xydias EM, Liasidi PN, Papageorgouli D, Tsakos E, Gouliopoulos N, Thanasas I, Daponte A, Ziogas AC. Three-dimensional transvaginal ultrasound versus MRI in the diagnosis and classification of congenital uterine anomalies: A systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2025 Aug;312:114560. doi: 10.1016/j.ejogrb.2025.114560. Epub 2025 Jul 2. PMID 40628082
- [Result] Tetlow RL, Richmond I, Manton DJ, Greenman J, Turnbull LW, Killick SR. Histological analysis of the uterine junctional zone as seen by transvaginal ultrasound. Ultrasound Obstet Gynecol. 1999 Sep;14(3):188-93. doi: 10.1046/j.1469-0705.1999.14030188.x. PMID 10550879
- [Result] Okaro E, Condous G, Khalid A, Timmerman D, Ameye L, Huffel SV, Bourne T. The use of ultrasound-based 'soft markers' for the prediction of pelvic pathology in women with chronic pelvic pain--can we reduce the need for laparoscopy? BJOG. 2006 Mar;113(3):251-6. doi: 10.1111/j.1471-0528.2006.00849.x. PMID 16487194
- [Result] Mukhopadhayay S, Bhattacharyya SK, Ganguly RP, Patra KK, Bhattacharya N, Barman SC. Comparative evaluation of perimenopausal abnormal uterine bleeding by transvaginal sonography, hysteroscopy and endometrial biopsy. J Indian Med Assoc. 2007 Nov;105(11):624, 626, 628 passim. PMID 18405088
- [Result] Babacan A, Gun I, Kizilaslan C, Ozden O, Muhcu M, Mungen E, Atay V. Comparison of transvaginal ultrasonography and hysteroscopy in the diagnosis of uterine pathologies. Int J Clin Exp Med. 2014 Mar 15;7(3):764-9. eCollection 2014. PMID 24753775
- [Result] Louis F, Lulla CP. Hysteroscopy is Superior to 3D Ultrasound in Gynecological Diagnosis. J Obstet Gynaecol India. 2020 Dec;70(6):447-461. doi: 10.1007/s13224-020-01384-8. Epub 2020 Dec 4. No abstract available. PMID 33417634
- [Result] Kolhe S. Management of abnormal uterine bleeding - focus on ambulatory hysteroscopy. Int J Womens Health. 2018 Mar 22;10:127-136. doi: 10.2147/IJWH.S98579. eCollection 2018. PMID 29606892
- [Result] Yasa C, Gungor Ugurlucan F. Approach to Abnormal Uterine Bleeding in Adolescents. J Clin Res Pediatr Endocrinol. 2020 Feb 6;12(Suppl 1):1-6. doi: 10.4274/jcrpe.galenos.2019.2019.S0200. PMID 32041387
- [Result] Pandey D, Kunamneni S, Inukollu PR, Su H. Establishing patterns on hysteroscopy in abnormal uterine bleeding (AUB). Gynecol Minim Invasive Ther. 2017 Oct-Dec;6(4):178-182. doi: 10.1016/j.gmit.2017.08.001. Epub 2017 Aug 26. PMID 30254909
- [Result] Ong CL. The current status of three-dimensional ultrasonography in gynaecology. Ultrasonography. 2016 Jan;35(1):13-24. doi: 10.14366/usg.15043. Epub 2015 Sep 25. PMID 26537304
- [Result] Turkgeldi E, Urman B, Ata B. Role of Three-Dimensional Ultrasound in Gynecology. J Obstet Gynaecol India. 2015 May;65(3):146-54. doi: 10.1007/s13224-014-0635-z. Epub 2014 Nov 8. PMID 26085733
- [Result] Wang L, Quan S, Bai E, Yang X. Analysis of clinical data of different endometrial pathological types in perimenopausal women with abnormal uterine bleeding. Front Oncol. 2024 Feb 29;14:1370681. doi: 10.3389/fonc.2024.1370681. eCollection 2024. PMID 38487719
- [Result] Dreisler E, Frandsen CS, Ulrich L. Perimenopausal abnormal uterine bleeding. Maturitas. 2024 Jun;184:107944. doi: 10.1016/j.maturitas.2024.107944. Epub 2024 Feb 22. PMID 38412750